CLINICAL TRIAL: NCT03311750
Title: Single-arm Phase II Study of Panitumumab Rechallenge in Combination With Oxaliplatin or Irinotecan-based Chemotherapy in Patients With RAS Wild Type Advanced Colorectal Cancer.
Brief Title: Anti-EGFR Therapy Rechallenge in Combination With Chemotherapy in Patients With Advanced Colorectal Cancer
Acronym: A-REPEAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: It was considered that the recruitment of the remaining 10 patients required of the trial will not be possible soon.
Sponsor: Hellenic Cooperative Oncology Group (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE6B/16; 2016-003644-37 (EudraCT Number)
Record Dates: First submitted 2017-10-02; First posted 2017-10-17 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Advanced Colorectal Cancer
MeSH Terms: interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Panitumumab (Experimental): On day 1 of each cycle patients will receive panitumumab followed by 5-fluorouracil and leucovorin in combination with either irinotecan (FOLFIRI regimen) or oxaliplatin (FOLFOX regimen) or followed by irinotecan monotherapy. This treatment will be repeated every 2 weeks for FOLFIRI and FOLFOX regimens and every 3 weeks for irinotecan monotherapy.
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab — 6 mg/Kg will be administered intravenous over 1 hour on Day 1 every 2 weeks or 9 mg/Kg every 3 weeks.
  Other Names: Vectibix

SUMMARY:
A-REPEAT (Anti-Epidermal Growth Factor Receptor -EGFR- rechallenge and plasma genotyping of patients with advanced colorectal tumors) is a Greek, investigator-initiated, single arm open-label phase II study of anti-EGFR therapy rechallenge in combination with chemotherapy in patients with advanced colorectal cancer. Patients with a metastatic, histologically proven colorectal carcinoma RAS wild type will be treated with a combination of panitumumab and third-line irinotecan-based or oxaliplatin-based chemotherapy (FOLFOX,FOLFIRI or irinotecan monotherapy).

DETAILED DESCRIPTION:
Few clinical studies have evaluated the role of anti-EGFR therapy rechallenge in metastatic colorectal cancer patients and there is no prospective clinical trial assessing the activity of treatment rechallenge with panitumumab-based therapy after initial progression. This study aims at exploring the concept of evolution and expansion of RAS wild type clones in order to restore sensitivity of the tumor to prior anti-EGFR therapy after a time interval in which a different, non-anti-EGFR second-line therapy is administered. Based on aforementioned data, it is hypothesized that rescue through rechallenge with panitumumab-based third-line therapy combined with chemotherapy could be associated with further response and clinical benefit. A significant component of the proposed prospective trial is exploratory translational: cell free plasma and platelet-based genotyping for genetic mutations in different time points will be undertaken in order to study the genetic composition of the metastatic tumour at initiation of and at progression through, anti-EGFR rechallenge therapy.

Primary endpoint will be to evaluate the efficacy, in terms of overall response rate, of the addition of panitumumab rechallenge to standard third-line irinotecan-based or oxaliplatin-based chemotherapy in patients with metastatic colorectal cancer initially treated with, and benefiting from, first line irinotecan-based or oxaliplatin-based chemotherapy combined with an anti-EGFR monoclonal antibody, followed by second line chemotherapy not containing anti-EGFR agents.

Exploratory endpoints include to identify, in the context of translational research, tumour tissue and blood-based biomarkers with prognostic/predictive significance in patients with metastatic colorectal cancer treated with rechallenge panitumumab in combination with standard third-line irinotecan-based or oxaliplatin-based chemotherapy, who were initially treated with, and benefiting from, first line irinotecan-based or oxaliplatin-based chemotherapy combined with an anti-EGFR monoclonal antibody, followed by second line chemotherapy not containing anti-EGFR agent.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent, and willing and able to comply with protocol requirements,
* Histologically proven adenocarcinoma of the colon and/or rectum,
* Metastatic disease confirmed clinically/radiologically,
* Patients with Formalin-Fixed, Paraffin-Embedded tissue RAS wild type colorectal cancer at diagnosis, who had initial clinical benefit [complete response, partial response or stable disease] during first line irinotecan-based or oxaliplatin-based chemotherapy in combination with cetuximab or panitumumab,
* First- line treatment duration (FOLFIRI, FOLFOX with anti-EGFR monoclonal antibody, of whom at least 2/3 of cases will have involved panitumumab) of at least 3 months,
* Second line therapy consisting of any chemotherapy (with or without Bevacizumab) definitely without anti-EGFR therapy of at least 2 months, followed by disease progression,
* Eligible third line regimens include FOLFIRI or Irinotecan or FOLFOX, according to standard practice and approved indications. It is required that the third line regimen used will be different from the second line and similar to the first line regimen,
* At least one measurable or evaluable lesion as assessed by computed tomography scan or Magnetic Resonance Imaging according to RECIST version 1.1,
* First course of treatment planned less than 1 week (7 days) after registration,
* Age ≥18 years,
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2,
* Adequate hematological status: neutrophils (ANC) ≥1.5x109/L; platelets ≥100x109/L; haemoglobin ≥9g/dL,
* Adequate renal function: serum creatinine level <1.5 mg/dL or Glomelular Filtration Rate (GFR) >50mL/min by Cockroft/Gault formula,
* Adequate liver function: serum bilirubin ≤1.5 x upper normal limit (ULN), alkaline phosphatase, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) <5xULN,
* Regular follow up feasible.
* For female patients of childbearing potential, negative serum or urine pregnancy test within 1 week (7 days) prior of starting study treatment
* Female patients must commit to using reliable and appropriate methods of contraception until at least three months after the end of study treatment (when applicable). Male patients with a partner of childbearing potential must agree to use contraception in addition to having their partner use another contraceptive method during the trial,
* Archival tumor tissue is required for exploratory research at enrolment,
* Ability to undergo plasma sampling during the therapy course.

Exclusion Criteria:

* Presence of central nervous system metastasis unless adequately treated (e.g. non irradiated central nervous system metastasis, seizures not controlled with standard medical therapy constitute non-eligibility criteria),
* Active infection (ie, body temperature ≥38°C due to infection),
* Intestinal obstruction, pulmonary fibrosis or interstitial pneumonitis, renal failure, liver failure, or cerebrovascular disorder,
* Uncontrolled diabetes,
* Myocardial infarction within the last 6 months, severe/unstable angina, symptomatic congestive heart failure New York Heart Association class III or IV,
* Known human immunodeficiency virus or acquired immunodeficiency syndrome-related illness, or hepatitis B or C,
* Autoimmune disorders or history of organ transplantation that require immunosuppressive therapy,
* Other concomitant or previous malignancy, except: i/ adequately treated in-situ carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer in complete remission for >5 years,
* Major surgery or traumatic injury within the last 28 days,
* Pregnant or breastfeeding women,
* Patients with known allergy to any excipients to study drugs,
* Other serious and uncontrolled chronic non-malignant disease,
* Known dihydropyrimidine dehydrogenase deficiency,
* Palliative radiation therapy within 4 weeks prior to registration,
* Life expectancy less than 12 weeks in the opinion of the Investigator,
* Treatment with any other investigational medicinal product within 28 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of overall response rate of the addition of panitumumab rechallenge to standard third-line therapy | At baseline, every 8 weeks with a 2-week tumor evaluation window through study completion, an average of 30 months.
  Evaluation of efficacy of overall response rate, of the addition of panitumumab rechallenge to standard third-line irinotecan-based or oxaliplatin-based chemotherapy in patients with metastatic colorectal cancer initially treated with, and benefiting from, first line irinotecan-based or oxaliplatin-based chemotherapy combined with an anti-EGFR monoclonal antibody, followed by second line chemotherapy not containing anti-EGFR agents.

SECONDARY OUTCOMES:
Evaluation of overall response rate by RAS status | At baseline, every 8 weeks with a 2-week tumor evaluation window through study completion, an average of 30 months.
  Overall response rate will be calculated separately for RAS mutant and wild type patients.Overall response rate is defined as the proportion of patients with confirmed complete response or partial response, as the best overall response to treatment, based on Response Evaluation Criteria in Solid Tumors version 1.1 guidelines
Evaluation of Progression Free Survival | From study entry to disease progression or death due to any cause assessed up to 30 months
Evaluation of Overall Survival | From study entry until date of death due to any cause or last contact assessed up to 30 months
Evaluation of safety of the combination of standard 3rd-line irinotecan-based or oxaliplatin-based chemotherapy with panitumumab rechallenge. | Per cycle (each cycle is repeated every 2 weeks for FOLFIRI and FOLFOX regimens and every 3 weeks for irinotecan monotherapy) assessed up to 30 months.
Mutation status of KRAS gene | At baseline
Mutation status of NRAS gene | At baseline
Next generation sequencing performed on plasma cell-free DNA. | At baseline, at cycle 3 or 4 (each cycle is repeated every 2 weeks for FOLFIRI and FOLFOX regimens and every 3 weeks for irinotecan monotherapy) and at progressive disease assessed up to 30 months
Mutations analysis on platelet-resorbed tumour RNA (with Real-time PCR) in Codon 12 of KRAS gene mutations | At baseline, at cycle 3 or 4 (each cycle is repeated every 2 weeks for FOLFIRI and FOLFOX regimens and every 3 weeks for irinotecan monotherapy) and at progressive disease assessed up to 30 months
Mutations analysis on platelet-resorbed tumour RNA (with Real-time PCR) in Codon 61 of KRAS gene mutations | At baseline, at cycle 3 or 4 (each cycle is repeated every 2 weeks for FOLFIRI and FOLFOX regimens and every 3 weeks for irinotecan monotherapy) and at progressive disease assessed up to 30 months
Mutations analysis on platelet-resorbed tumour RNA (with Real-time PCR) in exon 15 of BRAF gene mutations | At baseline, at cycle 3 or 4 (each cycle is repeated every 2 weeks for FOLFIRI and FOLFOX regimens and every 3 weeks for irinotecan monotherapy) and at progressive disease assessed up to 30 months
Mutations analysis on platelet-resorbed tumour RNA (with Real-time PCR) in Codon 12 of NRAS gene mutations | At baseline, at cycle 3 or 4 (each cycle is repeated every 2 weeks for FOLFIRI and FOLFOX regimens and every 3 weeks for irinotecan monotherapy) and at progressive disease assessed up to 30 months
Mutations analysis on platelet-resorbed tumour RNA (with Real-time PCR) in Codon 61 of NRAS gene mutations | At baseline, at cycle 3 or 4 (each cycle is repeated every 2 weeks for FOLFIRI and FOLFOX regimens and every 3 weeks for irinotecan monotherapy) and at progressive disease assessed up to 30 months
Mutations analysis on platelet-resorbed tumour RNA (with Real-time PCR) in exon 20 of PIK3CA gene mutations | At baseline, at cycle 3 or 4 (each cycle is repeated every 2 weeks for FOLFIRI and FOLFOX regimens and every 3 weeks for irinotecan monotherapy) and at progressive disease assessed up to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Sgouros, MD, Principal Investigator — 3rd Department of Medical Oncology,Agii Anargiri Cancer Hospital
Locations (8):
- Bank Of Cyprus Oncology Centre, Stróvolos, Nicosia, Cyprus
- Greece (7):
  - "Attikon" University Hospital, Chaïdári, Athens
  - University Hospital of Heraklion, Heraklion, Crete
  - Ioannina University Hospital, Ioannina, Ioannina
  - Agii Anargiri Cancer Hospital, Athens, Kalyftaki, Nea Kifisia
  - Metropolitan Hospital, Athens, Neo Faliro
  - University Hospital of Patra, Rio, Patra
  - Euromedica General Clinic of Thessaloniki, Thessaloniki, Thessaloniki